CLINICAL TRIAL: NCT04649255
Title: Liquid Embolization of Arterial Hemorrhages in the Peripheral Vasculature: The LAVA Study
Brief Title: Treatment of Peripheral Arterial Hemorrhage With Lava LES (The LAVA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlackSwan Vascular, Inc. (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR-00913-01.A
Record Dates: First submitted 2020-11-23; First posted 2020-12-02 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Arterial Hemorrhage
Keywords: Peripheral Arterial Hemorrhage; Embolic Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Lava LES (Experimental)
  Interventions: Device: Liquid Embolic

INTERVENTIONS:
Device: Liquid Embolic — Lava Liquid Embolic System (LES)

SUMMARY:
To evaluate the safety and effectiveness of the Lava LES for the embolic treatment of arterial hemorrhage in the peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Active arterial bleeding in the peripheral vasculature, documented on a suitable imaging study;
* Subject or subject's legally authorized representative is able and authorized to provide written informed consent for the procedure and the study;
* Subject is willing and able to comply with the specified follow-up evaluation schedule;
* Life expectancy >30 days;
* No prior embolization in the target territory.

Exclusion Criteria:

* Pregnancy or breast feeding. A woman who, in the Investigator's opinion, is of child-bearing potential must have a negative pregnancy test within 7 days before the index procedure;
* Coexisting signs of peritonitis or other active infection;
* Participation in an investigational study of a new drug, biologic or device that has not reached its primary endpoint at the time of study screening;
* Uncorrectable coagulopathies such as thrombocytopenia <40,000/ μL, international normalization ratio (INR) >2.0;
* Contraindication to angiography or catheterization, including untreatable allergy to iodinated contrast media;
* Anatomic arterial unsuitability such that, in the Investigator's opinion, the delivery catheter cannot gain access to the selected position for safe and intended embolization;
* Known allergy or other contraindication to any components of Lava LES including dimethyl sulfoxide (DMSO);
* More than 4 Target Lesions will require embolization, in the Investigator's opinion after performance of diagnostic angiography or another suitable imaging study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Arslan, MD, Principal Investigator — Rush University Medical Center; Mahmood Razavi, MD, Principal Investigator — St. Joseph Heart and Vascular Center
Locations (9):
- United States (9):
  - University of California, Irvine, California
  - University of Southern California, Los Angeles, California
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Albany University Medical Center, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject screening commenced on April 14, 2021 with the first subject enrolled on April 14, 2021. 160 subjects were screened at 20 investigational sites in the United States of America with no more than 25 subjects enrolled at any single site. 113 subjects were enrolled (successful arterial access established to the target lesion) at 19 sites in the Intent to treat (ITT) population.
Period: Overall Study
Arm/Group | Lava LES
Started | 113
Completed | 103
Not Completed | 10
Not completed — Death | 9
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lava LES
Number analyzed (Participants) | 113
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [18.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Out of the overall 113 participants, race data was available for 108 participants.
  Participants
    Asian: number analyzed (Participants) | 108
    Asian | 10
    Black or African-American: number analyzed (Participants) | 108
    Black or African-American | 16
    Native Hawaiian or other Pacific Islander: number analyzed (Participants) | 108
    Native Hawaiian or other Pacific Islander | 1
    White: number analyzed (Participants) | 108
    White | 63
    Other (Not otherwise specified): number analyzed (Participants) | 108
    Other (Not otherwise specified) | 18
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (6.88)
Target Bleed Territory - Upper GI [Count of Participants; unit: Participants]
  Upper GI | 11
  Lower GI | 10
  Non-GI Visceral | 41
  Extremity | 8
  Other (Not otherwise specified) | 43
Etiology of Bleeding [Count of Participants; unit: Participants]
  Traumatic, non-iatrogenic | 32
  Iatrogenic | 29
  Ulcer | 5
  Benign Neoplasm | 1
  Malignant Neoplasm | 5
  Mallory Weiss Tear | 0
  Congenital Vascular Lesion | 0
  Unknown | 6
  Other (Not otherwise specified) | 35
Currently Taking Antiplatelet Agents [Count of Participants; unit: Participants] — Population: Difference between number analyzed and overall was due to missing data.
  Participants
    number analyzed (Participants) | 96
    (all) | 9
Currently Taking Anticoagulant Agents [Count of Participants; unit: Participants] — Population: Difference between number analyzed and overall was due to missing data.
  Participants
    number analyzed (Participants) | 90
    (all) | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite of Freedom From Major Adverse Events (MAEs)
Description: A composite of freedom from 30-day MAEs include ischemia or infarction of the target territory, non-target embolization, allergic reactions to Lava, catheter breakage, and catheter entrapment defined as the inability to withdraw a catheter from adherence to Lava.
Time Frame: 30 Days
Population: Analysis based on the intent-to-treat (ITT) population with valid assessment. The baseline number of subjects was 113 but only 101 subjects were administered the assigned intervention (Lava LES), thus 101 subjects were evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lava LES
Number analyzed (Participants) | 101
percentage of participants | 100 [96.4 to 100]
Statistical Analysis 1: Comparison: Lava LES; Descriptive assessment; H0: Ps ≤ PGS, versus HA: PS > PGS, where where Ps is the population primary safety success rate in the Test group and PGS is the safety performance goal of 82%; Test type: Other; p < 0.025, One-sided exact binomial test; Exact binomial one-sided lower 97.5% CI for performance goal test >72% for primary effectiveness and >82% for primary safety; Exact binomial = 96.4, 95% CI 2-sided [96.4 to 100]

2. Primary Outcome: Percentage of Lesions to Achieve Clinical Success
Description: Defined as absence of bleeding from the target lesion after embolization with the Lava LES, without the need for emergency surgery, re-embolization, or other target lesion reinterventions.
Time Frame: 30 days
Population: Analysis based on the intent-to-treat (ITT) population with valid assessment.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: number of lesions
Arm/Group | Lava LES
Number analyzed (Participants) | 113
Number analyzed (number of lesions) | 141
percentage of lesions | 94.3 [89.1 to 97.5]
Statistical Analysis 1: Comparison: Lava LES; Descriptive assessment; H0: PE ≤ PGE, versus HA: PE > PGE, where PE is the proportion of target lesions with clinical success and PGE is the effectiveness performance goal of 72%; Test type: Other; p < 0.025, One-sided exact binomial test; [statistical method as in outcome 1, analysis 1]; Exact binomial = 89.1, 95% CI 2-sided [89.1 to 97.5]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks.
Description: Note: The primary and secondary safety endpoints were the major AEs at 30 days, and All-Cause Mortality through 30 days follow-up, hence the difference in the denominators.
  The denominator for total number of treated participants was 113, which was used for all general AE and SAE tables.
  The denominator for All-Cause Mortality was actually 109 because 4 participants were excluded due to exiting the study before the 30-day follow-up visit, without death.
Arm/Group | Lava LES
All-Cause Mortality (participants affected / at risk) | 9/113
Serious Adverse Events (participants affected / at risk) | 49/113
Other Adverse Events (participants affected / at risk) | 92/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lava LES (N=113)
Anaemia (Blood and lymphatic system disorders) | 3
Chronic myeloid leukaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac arrest (Cardiac disorders) | 1
Chest pain (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Small intestinal perforation (Gastrointestinal disorders) | 1
Death (General disorders) | 3
Flank pain (General disorders) | 2
Cholangitis infective (Hepatobiliary disorders) | 1
Gallbladder rupture (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 4
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2
Acute respiratory failure (Metabolism and nutrition disorders) | 1
Respiratory failure (Metabolism and nutrition disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Colectomy (Surgical and medical procedures) | 1
Cardiogenic shock (Vascular disorders) | 1
Epistaxis (Vascular disorders) | 1
Extravasation blood (Vascular disorders) | 3
Haematoma infection (Vascular disorders) | 1
Hepatic haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Retroperitoneal haematoma (Vascular disorders) | 1
Septic shock (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lava LES (N=113)
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Ascites (Cardiac disorders) | 2
Dizziness (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 4
Deafness unilateral (Ear and labyrinth disorders) | 1
Hypoglycaemia (Endocrine disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain lower (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenitis (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Omental haemorrhage (Gastrointestinal disorders) | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Cachexia (General disorders) | 1
Oedema (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 4
Bile duct stenosis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Haemangioma of liver (Hepatobiliary disorders) | 1
Infusion related reaction (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Klebsiella test positive (Investigations) | 1
White blood cell count increased (Investigations) | 1
Acidosis (Investigations) | 1
Dehydration (Investigations) | 1
Hyperkalaemia (Investigations) | 1
Lactic acidosis (Investigations) | 1
Tumour lysis syndrome (Investigations) | 1
Arthralgia (Investigations) | 3
Back pain (Investigations) | 2
Groin pain (Investigations) | 1
Inguinal mass (Investigations) | 1
Joint swelling (Investigations) | 1
Pain in extremity (Investigations) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Anuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
Urosepsis (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Hypoaesthesia (Skin and subcutaneous tissue disorders) | 1
Paraesthesia (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Dialysis device insertion (Surgical and medical procedures) | 1
Nephrostomy (Surgical and medical procedures) | 1
Pancreatic duct drainage (Surgical and medical procedures) | 1
Transfusion (Surgical and medical procedures) | 1
Contusion (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hepatic haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Renal infarct (Vascular disorders) | 1
Splenic haemorrhage (Vascular disorders) | 1
Splenic infarction (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04649255/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04649255/SAP_003.pdf